CLINICAL TRIAL: NCT03846479
Title: Itacitinib Monotherapy for Low Risk Graft-vs-Host Disease
Brief Title: Itacitinib for Low Risk GVHD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: John Levine (Other)
Responsible Party: Sponsor-Investigator, John Levine, Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 18-1684
Record Dates: First submitted 2019-02-17; First posted 2019-02-19 (Actual); Results first posted 2023-02-06 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Low Risk Acute Graft-versus-host Disease; Graft-versus-host-disease; GVHD
Keywords: Graft-versus-host disease; Itacitinib
MeSH Terms: conditions — Graft vs Host Disease | interventions — itacitinib

STUDY DESIGN:
Intervention Model Description: Open label, single arm, non-inferiority study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Itacitinib (Experimental): Itacitinib 200 mg administered orally daily
  Interventions: Drug: Itacitinib

INTERVENTIONS:
Drug: Itacitinib — for up to 56 days
  Other Names: INCB389110

SUMMARY:
Graft-versus-host disease (GVHD) is treated with high doses of systemic steroids which can lead to serious complications. A new blood test can identify patients whose GVHD is most likely to respond to well to treatment (low risk GVHD). This study will test whether patients with low risk GVHD can be successfully treated without steroids. Patients who participate with this study will be treated with itacitinib instead of steroids. Itacitinib is an experimental drug with an excellent safety record and appears to have activity as a GVHD treatment.

DETAILED DESCRIPTION:
Patients with newly diagnosed low risk acute GVHD defined as Minnesota standard risk based on symptoms and Ann Arbor 1 GVHD based on biomarkers were eligible if they met all other eligible criteria (see eligibility criteria below). Enrolled patients were required to start treatment within 4 days of confirmation of Ann Arbor 1 status. Treatment consisted of itacitinib 200 mg daily for 28 days. Patients with a clinical response on day 28 were eligible for a second 28 day cycle of itacitinib 200 mg daily. Missed doses could be made up by extending the treatment duration for up to 2 additional weeks. Medications given for GVHD prophylaxis and topical treatments for GVHD were allowed. Supportive care was provided according to institutional standards. Itacitinib was permanently discontinued after any of the following:

administration of 56 doses of itacitinib or initiation of systemic corticosteroids or any other systemic treatment for GVHD or patient withdrawal from the study or general or specific changes in the patient's condition render the patient unacceptable for further treatment in the judgment of the investigator OR ten weeks elapsed since the first dose of itacitinib.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed GVHD that meets criteria for Minnesota standard risk
* Ann Arbor 1 GVHD by biomarkers
* GVHD not previously treated systemically (topical therapies and non-absorbed steroids are allowed)
* Any donor type, HLA-match, conditioning regimen is acceptable
* Age 12 - 75 years (children <18 years must also weigh 50 kg or more)
* Patients must be engrafted post-transplant (ANC >500/μL and platelet count >20,000). Use of growth factor supplementation to maintain neutrophil count is allowed.
* Direct bilirubin must be <2 mg/dL unless the elevation is known to be due to Gilbert syndrome within 3 days prior to enrollment.
* ALT/SGPT and AST/SGOT must be <5x the upper limit of the normal range within 3 days prior to enrollment.
* Signed and dated written informed consent obtained from patient or legal representative.

Exclusion Criteria:

* Patients currently being treated with any JAK inhibitor including ruxolitinib
* Relapsed, progressing, or persistent malignancy requiring withdrawal of systemic immune suppression
* Patients with uncontrolled infection (i.e., progressive symptoms related to infection despite treatment or persistently positive microbiological cultures despite treatment or any other evidence of severe sepsis)
* Severe organ dysfunction including requirement for dialysis, mechanical ventilation or oxygen supplementation exceeding 40% FiO2 within 7 days of enrollment.
* Creatinine clearance or estimated glomerular filtration rate <30 ml/min as calculated by institutional practice (e.g., Cockcroft-Gault equation, CKD-EPI equation, etc)
* A clinical presentation resembling de novo chronic GVHD or overlap syndrome developing before or present at the time of enrollment
* Patients receiving corticosteroids >10 mg/day prednisone (or other steroid equivalent) for any indication within 7 days before the onset of acute GVHD except for adrenal insufficiency or premedication for transfusions/IV meds
* Patients who are pregnant
* Patients receiving investigational agents within 30 days of enrollment. However, the Principal Investigator (PI) may approve prior use of an investigational agent if the agent is not expected to interfere with the safety or the efficacy of itacitinib
* History of allergic reaction to itacitinib or any JAK inhibitor

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2021-05-07 (Actual); Study Completion 2022-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Levine, MD, MS, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (14):
- United States (14):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Emory University, Atlanta, Georgia
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - University of Kansas Cancer Center, Fairway, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - The Mount Sinai Hospital, New York, New York
  - Ohio State University, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pennsylvania, Abramson Cancer Center, Philadelphia, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Etra A, Capellini A, Alousi A, Al Malki MM, Choe H, DeFilipp Z, Hogan WJ, Kitko CL, Ayuk F, Baez J, Gandhi I, Kasikis S, Gleich S, Hexner E, Hoepting M, Kapoor U, Kowalyk S, Kwon D, Langston A, Mielcarek M, Morales G, Ozbek U, Qayed M, Reshef R, Rosler W, Spyrou N, Young R, Chen YB, Ferrara JLM, Levine JE. Effective treatment of low-risk acute GVHD with itacitinib monotherapy. Blood. 2023 Feb 2;141(5):481-489. doi: 10.1182/blood.2022017442. PMID 36095841

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Risk GVHD Patients Treated: Itacitinib 200 mg administered orally daily for 28 days, with a second 28 day cycle allowed for responding patients.
Period: Overall Study
Arm/Group | Low Risk GVHD Patients Treated
Started | 70
Completed | 61
Not Completed | 9
Not completed — Death | 8
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Low Risk GVHD Patients Treated
Number analyzed (Participants) | 70
Age, Continuous [Median (Full Range); unit: years] | 60 [15 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 59
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 57
  More than one race | 0
  Unknown or Not Reported | 4
Diagnosis [Count of Participants; unit: Participants]
  Acute Leukemia | 32
  MDS, myelodysplastic syndrome; MPN, myeloproliferative neoplasm (MDS/MPN) | 29
  Lymphoma | 6
  Non-Malignant | 3
Donor [Count of Participants; unit: Participants]
  Matched related | 13
  Matched unrelated | 37
  Mismatched related | 15
  Mismatched unrelated | 5
Conditioning Regimen [Count of Participants; unit: Participants] — Pre-transplant chemotherapy regimen categorized as either myeloablative or reduced/non-myeloablative intensity.
  Participants
    Myeloablative | 33
    Reduced/Non-Myeloablative | 37
Anti-Thymocyte Globulin (ATG) [Count of Participants; unit: Participants]
  Yes | 9
  No | 61
GVHD Prophylaxis [Count of Participants; unit: Participants] — CNI = calcineurin inhibitor
  MTX = Methotrexate
  MMF = mycophenolate
  Participants
    CNI/MTX (+/- Other) | 24
    CNI/MMF (+/- Other) | 7
    CNI/sirolimus | 2
    Cyclophosphamide based | 35
    T Cell Depletion | 2
    Other | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Achieve CR or PR by Day 28 of Treatment
Description: Number of patients who achieve CR or PR by day 28 of treatment with itacitinib without the addition of any other systemic GVHD treatment including steroids.
  Complete Response (CR): All evaluable organs (skin, liver, GI tract) stage 0. For a response to be scored as CR on day 28, the patient must be in CR on that day and have had no intervening additional GVHD therapy.
  Partial Response (PR): An improvement in one or more organ involved with GVHD symptoms without worsening in others. For a response to be scored as PR on day 28, the patient must be in PR on that day and have had no intervening additional GVHD therapy.
Time Frame: Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Low Risk GVHD Patients Treated
Number analyzed (Participants) | 70
Participants | 62

2. Primary Outcome: Number of Participants Who Developed Steroid Refractory GVHD
Description: Number of participants who developed steroid refractory GVHD within 28 days of starting steroids. Steroid-refractory GVHD (defined as GVHD that worsens (increase by one or more grade) after 3 days, or fails to respond to treatment within 7 days (for GVHD grade III) or 14 days (for GVHD grade II) or 2nd line therapy beyond systemic steroid treatment is begun within 28 days of starting steroids.
Time Frame: Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Low Risk GVHD Patients Treated
Number analyzed (Participants) | 70
Participants | 1

3. Secondary Outcome: Number of Participants With Serious Infectious
Description: Number of participants who developed serious infections by day 90. Serious infectious complications is defined as any viral and bacterial infections requiring treatment and proven fungal infections.
Time Frame: Day 90
Measure: Count of Participants; unit: Participants
Arm/Group | Low Risk GVHD Patients Treated
Number analyzed (Participants) | 70
Participants | 19

4. Secondary Outcome: Number of Participants Alive at 6 Months and 1 Year
Description: Number of overall survival (OS), defined as the duration from the date of diagnosis to death or last follow-up, with no restriction on the cause of death.
Time Frame: 6 months and 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Low Risk GVHD Patients Treated
Number analyzed (Participants) | 70
Participants
  6 months | 66
  1 year | 62

5. Secondary Outcome: Number of Participants With Non-relapse Mortality (NRM)
Description: Number of participants with non-relapse mortality (NRM) at 6 months and 1 year
Time Frame: 6 months and 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Low Risk GVHD Patients Treated
Number analyzed (Participants) | 70
Participants
  6 months | 2
  1 year | 3

6. Secondary Outcome: Number of Participants Who Relapsed
Description: Number of participants who relapsed by 6 months and by 1 year
Time Frame: 6 months and 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Low Risk GVHD Patients Treated
Number analyzed (Participants) | 70
Participants
  6 months | 8
  1 year | 12

7. Secondary Outcome: Number of Participants Who Developed Chronic GVHD
Description: Number of participants who developed chronic GVHD requiring systemic treatment at 1 year
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Low Risk GVHD Patients Treated
Number analyzed (Participants) | 70
Participants | 18

8. Secondary Outcome: Cumulative Steroid Dose
Description: Cumulative steroid dose (over 4 weeks) in patients who receive steroids as second line therapy
Time Frame: Day 28
Measure: Mean (Standard Error); unit: mg/kg
Arm/Group | Low Risk GVHD Patients Treated
Number analyzed (Participants) | 70
mg/kg | 1.9 (0.6)

ADVERSE EVENTS:
Time Frame: 90 days for Adverse Events 1 year for All-Cause Mortality
Arm/Group | Low Risk GVHD Patients Treated
All-Cause Mortality (participants affected / at risk) | 8/70
Serious Adverse Events (participants affected / at risk) | 23/70
Other Adverse Events (participants affected / at risk) | 34/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Risk GVHD Patients Treated (N=70)
Fever (General disorders) | 3
Dysuria (Renal and urinary disorders) | 1
Subarachnoid Hemorrhage (Injury, poisoning and procedural complications) | 1
Adenovirus Hemorrhagic Cystitis (Infections and infestations) | 1
Acute Kidney Injury (Renal and urinary disorders) | 1
Syncope (Nervous system disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
GVHD (Immune system disorders) | 4
Blood Bilirubin Increased (Investigations) | 1
Hypertension (Vascular disorders) | 1
Relapse (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
C. Difficile Infection (Infections and infestations) | 3
SARS-CoV-2 Infection (Infections and infestations) | 1
EBV Infection (Infections and infestations) | 1
BK Cystitis (Infections and infestations) | 2
Sepsis (Infections and infestations) | 3
Catheter Related Infection (Infections and infestations) | 4
Bacteremia (Infections and infestations) | 2
Upper Respiratory Infection (Infections and infestations) | 1
Lung Infection (Infections and infestations) | 1
CMV Viremia (Infections and infestations) | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 2
Suicidal Ideation (Psychiatric disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Risk GVHD Patients Treated (N=70)
Anemia (Blood and lymphatic system disorders) | 14
Syncope (Nervous system disorders) | 1
Hypertension (Vascular disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 1
White Blood Cell Decreased (Investigations) | 11
Lymphocyte Count Decreased (Investigations) | 2
Neutrophil Count Decreased (Investigations) | 11
Reversible Posterior Leukoencephalopathy Syndrome (Nervous system disorders) | 1
Platelet Count Decreased (Investigations) | 13
Thrombotic Microangiopathy (Vascular disorders) | 1
Headache (Nervous system disorders) | 1
Alanine Aminotransferase Increased (Investigations) | 5
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1
Urinary Tract Infection (Infections and infestations) | 1
CMV Infection (Infections and infestations) | 3
EBV Infection (Infections and infestations) | 1
Multifocal Pneumonia (Infections and infestations) | 1
Arthralgia and/or Myalgia (Musculoskeletal and connective tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-13): https://cdn.clinicaltrials.gov/large-docs/79/NCT03846479/Prot_SAP_000.pdf